CLINICAL TRIAL: NCT05461560
Title: Investigating the Effects of Seaweed Extract on Postprandial Blood Glucose Response to Sucrose in Healthy Subjects
Brief Title: Effects of Seaweed Extract on Blood Glucose Response to Sucrose
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Dublin (Other)
Responsible Party: Principal Investigator, Akristic, Assistant Professor, University College Dublin
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: LS-21-54
Record Dates: First submitted 2022-07-13; First posted 2022-07-18 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Glucose Intolerance; Diabetes Mellitus, Type 2; Healthy Diet; Postprandial Hyperglycemia
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2; Hyperglycemia | interventions — sodium lactobionate sucrose solution

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Sucrose solution (Sham Comparator): Participants will consume 50g of sucrose dissolved in 500 ml of tap water
  Interventions: Dietary Supplement: Sucrose solution
- Experimental: Seaweed extract in sucrose solution (Experimental): Participants will consume 50g of sucrose and 1g of seaweed extract dissolved in 500 ml of tap water
  Interventions: Dietary Supplement: Seaweed extract in sucrose solution

INTERVENTIONS:
Dietary Supplement: Sucrose solution — 50 g of sucrose dissolved in 500 ml of tap water
  Arms: Control: Sucrose solution
Dietary Supplement: Seaweed extract in sucrose solution — 1 g of seaweed extract in solution of 50 g of sucrose in 500 ml of tap water
  Arms: Experimental: Seaweed extract in sucrose solution

SUMMARY:
This study will examine the impact of the seaweed (Ascophyllum nodosum) extract on blood glucose levels after a sugary drink in healthy subjects.

The aim of this study is to investigate if the seaweed extract, when consumed with the sucrose, can lower blood glucose levels, compared to the raise after sucrose only, in healthy volunteers.

The study is designed as an acute, double-blind, randomised, controlled crossover trial in 16 healthy subjects. Participants will be asked to consume sucrose solution or sucrose solution with added seaweed extract.The effects on blood glucose levels will be determined over 2 hours after the consumption.

DETAILED DESCRIPTION:
Blood glucose levels after a meal rich in sugars depend, among other factors, on the activity of enzymes that digest sugar molecules to glucose. Epidemiological studies suggest that glucose levels after a meal higher than normal, present a great risk for the onset of cardiovascular diseases. Slowing the digestion of sugar through the inhibition of digestion enzymes have been demonstrated as a successful approach in preventing postprandial hyperglycaemia either with pharmacological agents (acarbose, miglitol) or natural dietary compounds.

We demonstrated, in preclinical in vitro experiments, the unique potential of tested seaweed extract to inhibit rat sucrase.

This study will examine the potential of the seaweed extract to modulate blood glucose levels after a sucrose drink in healthy subjects .

The aim of this study is to investigate if the seaweed extract, when consumed with sucrose, can lower blood glucose levels, compared to the raise after sucrose only.

The study is designed as an acute, double-blind, randomised, controlled crossover trial in 16 healthy subjects. Participants will be asked to consume sucrose solution or sucrose solution with added seaweed extract.The effects on blood glucose levels (in capillary blood) will be determined over 2 hours after the consumption. All participants will be characterized for the activity of salivary a-amylase

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years
* Healthy

Exclusion Criteria:

* Smoking
* Diagnosis of any chronic illness (including diabetes, hypertension, gastrointestinal diseases etc.)
* On long term prescribed medication (except contraceptives)
* Pregnant or lactating
* On a special diet or dietary regimen (for weight management or if regularly consuming fruit extract supplements)
* Allergy to fruits vegetables, pollen or seaweed.
* Unwillingness to follow dietary recommendations or record the diet during recommended period
* Donated blood 4 weeks before or intend to donate blood during the study or 4 weeks after the last study samples
* Participation in another research project in parallel which also involves dietary intervention (e.g. taking vitamin supplements) or requires sampling of blood

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-05 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in maximal incremental capillary blood glucose level (iCmax) between baseline and endpoint within the intervention group vs. control. | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes
  The incremental glucose levels will be determined for each time point (at 15, 30, 45, 60, 90, 120 minutes) as the change in capillary blood glucose levels after the consumption of seaweed extract in sucrose solution or sucrose solution, compared to the glucose levels before the consumption of test drinks (baseline value, t=0 minutes)

SECONDARY OUTCOMES:
Changes in area under the curve of incremental capillary blood glucose levels (iAUC) in the intervention group vs. control | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes
  The glucose iAUC will be determined from all incremental capillary blood glucose levels at the defined time points (0, 15, 30, 45, 60, 90, 120 minutes) after the consumption of test and control drinks based on trapezoid rule.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Food and Health Volunteer Suite; Science Center South, UCD, Dublin, Dublin 2, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Access to the data by a 3rd party will only be given through collaboration with one of the existing PIs. The data may be shared for other research projects, and in an anonymised form. Consent to share the data for such purposes is requested in the study consent form.
Supporting Information: Study Protocol